**Dated: April 30, 2024** 

#### INTRODUCTION

Root canal therapy (RCT) stands as the primary treatment modality for pulpal and periapical diseases <sup>[1]</sup>. An indispensable facet of Root canal therapy involves the meticulous processes of cleaning, shaping, and subsequent obturation of the root canal system, establishing a robust and impermeable seal <sup>[1,2]</sup>. The prognosis of Root canal therapy hinges upon various factors, including irrigation techniques and the technical proficiency of the root filling <sup>[3]</sup>.

Throughout its evolution, root canal irrigation has seen diverse methodologies employed to effectively disinfect the root canal space. Traditionally, techniques such as syringe irrigation and passive ultrasonic irrigation have been prevalent <sup>[4]</sup>. However, the introduction of ultrasonic activation irrigation systems has added a dynamic dimension, utilizing ultrasonic energy to augment irrigant flow and disrupt biofilms. Root canal irrigation plays a pivotal role in Endodontics, facilitating instrumentation through lubrication, removal of debris, microorganisms, smear layer, and preventing apical debris packing. Irrigants exert their effects through mechanical, chemical, and biological actions <sup>[5]</sup>.

Activated irrigation involves agitating and enhancing the flow of irrigants into the intricacies of the root canal system using mechanical or other energy forms. Unlike conventional irrigation, which relies solely on positive pressure and the viscosity of the irrigant for flow in the root canal system <sup>[5,6]</sup>, various mechanical irrigant activation systems are available. These include ultrasonic activation using high or low frequency (e.g., EndoActivator), continuous ultrasonic irrigation (CUI), special holding devices during ultrasonics like Nusstein's needle holding device, sonic energy (RispiSonic file), vibrations (Vibringe), passive ultrasonic irrigation (PUI-IrriSafe), and positive or negative pressure alternating devices (EndoVac, RinsEndo), or manual agitation of

**Dated:**April 30, 2024

the irrigant with high amplitude/frequency (MDA) <sup>[5-7]</sup>. The efficacy of irrigation depends on both the mode of delivery and the irrigant itself <sup>[5]</sup>.

The primary objective of root canal obturation is to achieve a fluid-tight seal to prevent future microbial contamination <sup>[8]</sup>. Obturation quality encompasses the length of the filling, density of the filling material, and the absence of voids <sup>[9]</sup>. The significance of achieving high-quality obturation cannot be overstated, directly impacting the prevention of microbial ingress and reinfection. Poor obturation may lead to treatment failure, necessitating retreatment and underscoring the importance of a comprehensive understanding of factors influencing obturation quality <sup>[10,11]</sup>.

Studies, such as the one by Chen S et al., have compared ultrasonic irrigation with syringe irrigation, revealing a higher incidence of lateral canal fill with ultrasonic irrigation (27% vs. 7% in syringe irrigation) [12]. Another study found no statistical difference in irrigant penetration in the main canal compared to control, passive ultrasonic irrigation, continuous ultrasonic irrigation, and easy clean groups [13]. Yet, a study demonstrated a significant difference in radiographic healing rates among three groups ( $\chi$ 2=12.29, p=0.05), with higher healing rates observed in the Passive ultrasonic irrigation group (36.8%) and Laser activated irrigation group (42.1%) compared to the Conventional Syringe irrigation group (10.5%) [14].

While many studies have explored outcomes such as post-operative pain, periapical healing, antibacterial efficacy, canal cleanliness, debridement efficacy, and delivery up to working length, limited research has directly compared obturation results between irrigation methods. Given the scarcity of data on this outcome and the direct impact of irrigation technique on the obturation quality and lateral canal fill, a systematic investigation is warranted. This study aims to address

Dated: April 30, 2024

this gap, contributing to the existing knowledge base and guiding clinicians in optimizing their endodontic procedures.

## **OBJECTIVE**

To compare the quality of Obturation and lateral canal fill (by sealer) during root canal treatment between two irrigation techniques—ultrasonic activated irrigation and non-ultrasonic conventional irrigation

### **OPERATIONAL DEFINITIONS**

### **Obturation Quality and Lateral canal fill**

It will include assessing the length of the root canal filling of main canals, evaluating the density of the filling material, determining the taper of root canal filling, and accessing the lateral canal fill by sealer by post- operative radiographs. The radiographs will be evaluated independently by two senior endodontists. A scoring system will be employed and each of three components will be given a score of 0 and 1 with higher scores indicating better obturation quality (Table 1, 2 and 3).

Dated:April 30, 2024

Table 1. Parameters used to evaluate and score the quality of RCTs

| Parameters | Criteria | Definition |
|---|---|---|
| Length of root canal filling | Adequate(=1) | Root filling ending ≤ 2 mm from the radio-graphic apex |
| | Inadequate(=0) | Overfilled: root filling extruded beyond the radio- graphic apex |
| | | Under-filled: root filling ≥2 mm from the radio- graphic apex |
| Density of root canal filling | Adequate(=1) | Correct density of filling material and no voids present in the root filling nor between root filling and root canal walls |
| | Inadequate(=0) | Low density of filling material and/or voids present in the root filling or between root filling and root canal walls |
| Taper of root canal filling | Adequate(=1) | Consistent taper from the coronal to the apical part of the |
| | | filling |

| Inadequate(=0) | No consistent taper from the |
|----------------|-----------------------------------|
| | coronal to the apical part of the |
| | filling |

### Table 2

## **T-Score**

| Score 3 | Obturated canals have all three qualities of ideal Obturation. Adequately filled (with in 2mm from radiographic apex). Smooth coronal apical taper. No voids |
|---|---|
| Score 2 | Obturated canals have any two qualities of ideal obturation. |
| Score 1 | Obturated canals have any one quality of ideal obturation. |
| Scorre o | Obturated canals have no quality of ideal obturations |

## Lateral canal:

A type of accessory canal located in the coronal or middle third of the root, usually extending horizontally from the main canal space.

Table 3

Parameters used to evaluate and score of lateral canal fill

| Score 1 | Adequete | Lateral canals were filled with |
|---------|-----------|---------------------------------|
| Score 0 | Inadequte | Lateral canals were not filled |

## **Non-Ultrasonic Conventional Irrigation**

Comparison of Quality of Obturation and Lateral Canal Fill (by Sealer): Ultrasonic Activated versus Non-Ultrasonic Conventional

Irrigation Techniques in Root Canal Treatment: A Randomized

**Controlled Trial** 

Dated: April 30, 2024

This group involves the application of irrigating solutions through syringes or irrigation needles during the root canal procedure. 5 ml of 3% sodium hypochlorite (NaOCl) solution will be

introduced into each canal via 5cc syringes.

**Ultrasonic Activated Irrigation Technique** 

This group involves the use of ultrasonic device to agitate and activate irrigating solutions within

the root canal.VAT-3 ultrasonic activator high frequency device (45KHz± 5kHz) [Refine] will be

used for this study and 3% sodium hypochlorite (NaOCl) solution will be used for irrigation.

**HYPOTHESIS** 

There is a difference in obturation quality and lateral canal fill between ultrasonic activated

irrigation results as compared to conventional irrigation technique in root canal treatment.

MATERIAL AND METHOD

STUDY DESIGN: Double Blinded Randomized Controlled Trial

STUDY SETTING: Operative Dentistry and Endodontics, Peshawar Dental College Peshawar

**DURATION OF STUDY:** Minimum six months, after the synopsis approval

**SAMPLING METHOD:** Non-Probability Consecutive Sampling

**SAMPLE SIZE:** Sample size is calculated using WHO calculator keeping 5% level of

significance, 90 % power of test, based on reference study, 27% of sampled population achieved

adequate obturation and lateral fill of canals in ultrasonic activated irrigation group as compared

Dated: April 30, 2024

to conventional non irrigation group which was 7% as shown in (table 4) [12]. Expected sample size is 59 participants in each group, total 118 patients.

Table 4 Comparison of lateral canal filling between the two groups

| Variable | Group S $(n = 30)$ | Group U $(n = 30)$ | $X^2$ | P value |
|---|---|---|---|---|
| Lateral canal root canal filling | 2 (7) | 8 (27) | 4.320 | 0.038 |

#### **SAMPLE SELECTION:**

#### **Inclusion Criteria:**

- Both male and female
- Age Group: Adults (18-70) Years
- Patients presenting with pain and sensitivity in the mandibular molars and are advised root canal treatment at our institute after examination and Xray

#### **Exclusion Criteria:**

- Teeth with complex root canal anatomy that may complicate the obturation process.
- Pregnancy
- Medically compromised patient including those with uncontrolled diabetes, cardiovascular diseases, immunodeficiency disorders, bleeding disorders, and severe respiratory diseases
- Patients who refused to participate in this study.

: Ultrasonic Activated versus Non-Ultrasonic Conventional Irrigation Techniques in Root Canal Treatment: A Randomized

## **Controlled Trial**

**Dated: April 30, 2024** 

### **DATA COLLECTION PROCEDURE:**

Ethical approval will be obtained from institutional research board of the hospital. Synopsis will be submitted for approval by CPSP. Once approved, patients will then be recruited from the endodontics department of Peshawar dental college who presents complaining of pain and sensitivity in the mandibular teeth and are candidates for RCT after dental examination and Xray teeth. Patients who get enrolled in the study will be screened for eligibility using the inclusion and exclusion criteria. This will be a double blinded study (the participant and the outcome assessor both will be kept blind). A written informed consent will be taken after explaining the purpose of study and will be given the opportunity to ask any questions they may have about the study. Demographic data regarding age, gender, will be noted. Similarly, additional information about the specific tooth under consideration, will be documented. After randomization into either the Non-Ultrasonic Conventional Irrigation or Ultrasonic Activated Irrigation group via block randomization, pre-operative radiographs will be taken to establish baseline conditions. A block size of 6 will be used to ensure equal allocation of participants into each group. The root canal treatment is then performed as per the assigned group, with conventional irrigation involving the use of syringes and 3% sodium hypochlorite solution and Tg Sealer for the Non-Ultrasonic Conventional Irrigation group, and the utilization of the VAT-3 ultrasonic activator high frequency device (45KHz± 5kHz) [Refine] for the Ultrasonic Activated Irrigation group and same solution of 3% sodium hypochlorite and Tg Sealer will be used. Post-operative radiographs will be obtained to assess the obturation quality and lateral canal fill. A detailed radiographic proforma

## : Ultrasonic Activated versus Non-Ultrasonic Conventional Irrigation Techniques in Root Canal Treatment: A Randomized

will be employed to evaluate the length, density, taper of the root canal filling, and lateral canal fill . Each of these components will be scored individually, and an overall

Obturation Quality Score is calculated by summing these scores. Care will be taken in the

## **Controlled Trial**

**Dated:**April 30, 2024

documentation of information so that information bias is reduced. All these information and other demographic will also be recorded into a predesigned proforma. Throughout the data collection process, the research team will maintain strict adherence to data protection and confidentiality guidelines.

#### DATA ANALYSIS PROCEDURE

Data will be analyzed by using statistical package for social sciences (SPSS) version 25. Mean  $\pm$  SD will be measured for numerical data i.e age of the patient. Normality of the data will be calculated by Shappiro Wilk test and Non-normal data will be presented as median (IQR). Frequencies and percentages will be measured for categorical data i.e gender, residence, socioeconomic status, type of tooth (Molars), side of tooth, teeth involved (Mandibular), and categorization of obturation score. Lateral canal Fill quality will be compared in each group by using the chi-square or fischer exact test, keeping p-value  $\leq 0.05$  as significant. Effect modifiers i.e age, gender, side of tooth and tooth involved will be controlled through stratification. Post stratification chi-square or fischer exact test will be performed by keeping the p-value  $\leq 0.05$  considered as significant.

## : Ultrasonic Activated versus Non-Ultrasonic Conventional Irrigation Techniques in Root Canal Treatment: A Randomized

### **REFERENCES:**

- 1. Karamifar K, Tondari A, Saghiri MA. Endodontic Periapical Lesion: An Overview on the Etiology, Diagnosis and Current Treatment Modalities. Eur Endod J. 2020;5(2):54-67.
- 2. Şanal Çikman A, Köse TE, Günaçar DN, Çene E, Arıcıoğlu B. Evaluation of endodontically treated teeth and related apical periodontitis using periapical and

## **Controlled Trial**

**Dated: April 30, 2024** 

endodontic status scale: Retrospective cone-beam computed tomography study. Aust Endod J. 2022;48(3):431-43.

- 3. Al-Manei KK. Radiographic Quality of Single vs. Multiple-Visit Root Canal Treatment Performed by Dental Students: A Case Control Study. Iran Endod J. 2018;13(2):149-54.
- 4. Dioguardi M, Gioia GD, Illuzzi G, Laneve E, Cocco A, Troiano G. Endodontic irrigants: Different methods to improve efficacy and related problems. Eur J Dent. 2018;12(3):45966
- 5. Susila A, Minu J. Activated Irrigation vs. Conventional non-activated Irrigation in Endodontics A Systematic Review. Eur Endod J. 2019;4(3):96-110.
- 6. Tonini R, Salvadori M, Audino E, Sauro S, Garo ML, Salgarello S. Irrigating Solutions and Activation Methods Used in Clinical Endodontics: A Systematic Review. Front Oral Health. 2022;3:e838043.
- 7. Middha M, Sangwan P, Tewari S, Duhan J. Effect of continuous ultrasonic irrigation on postoperative pain in mandibular molars with nonvital pulps:a randomized clinical trial. Int Endod J. 2017;50(6):522–30.

## : Ultrasonic Activated versus Non-Ultrasonic Conventional Irrigation Techniques in Root Canal Treatment: A Randomized

- 8. Kim SY, Jang YE, Kim BS, Pang EK, Shim K, Jin HR, et al. Effects of Ultrasonic Activation on Root Canal Filling Quality of Single-Cone Obturation with Calcium Silicate-Based Sealer. Materials (Basel). 2021;14(5):e1292.
- Al-Anesi MS, AlKhawlani MM, Alkheraif AA, Al-Basmi AA, Alhajj MN. An audit of root canal filling quality performed by undergraduate pre-clinical dental students, Yemen. BMC Med Educ. 2019;19(1):350

-Ultrasonic Conventional : A Randomized

## : Ultrasonic Activated versus Non Irrigation Techniques in Root Canal Treatment Controlled Trial

## **Dated:**April 30, 2024

- 10. Gulabivala K, Ng YL. Factors that affect the outcomes of root canal treatment and retreatment—A reframing of the principles. Int Endod J. 2023;56:82-115.
- 11. Zhang P, Yuan K, Jin Q, Zhao F, Huang Z. Presence of voids after three obturation techniques in band\_shaped isthmuses: a micro\_computed tomography study. BMC Oral Health. 2021;21(1):227-30.
- 12. Chen S, Liu J, Dong G, Peng B, Yang P, Chen Z, et al. Comparison between ultrasonic irrigation and syringe irrigation in clinical and laboratory studies. J Oral Sci. 2016;58(3):373-8.
- 13. Souza CC, Bueno CE, Kato AS, Limoeiro AG, Fontana CE, Pelegrine RA. Efficacy of passive ultrasonic irrigation, continuous ultrasonic irrigation versus irrigation with reciprocating activation device in penetration into main and simulated lateral canals. J Conserv Dent. 2019;22(2):155-9.
- 14. Verma A, Yadav RK, Tikku AP, Chandra A, Verma P, Bharti R, et al. A randomized controlled trial of endodontic treatment using ultrasonic irrigation and laser activated irrigation to evaluate healing in chronic apical periodontitis. J Clin Exp Dent. 202;12(9):e821-e9

# COMPARISION OF QUALITY OF OBTURATION AND LATERAL CANAL FILL (BY SEALER): ULTRASONIC ACTIVATED VERSUS NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUES IN ROOT CANAL TREATMENT:- A Randomized Controlled Trial

Dated: April 30, 2024

## **Data Collection Proforma**

| Participant Information: |
|---|
| Participant ID: |
| Age [years]: |
| Gender: [male / female] |
| Residenc [Rural / Urban]: |
| Socioeconomic status [Low / Moderate / High ]: |
| <ul> <li>Low = &lt;50K PKR monthly Household income</li> <li>Moderate = 50K to 150K PKR monthly household income</li> <li>High = &gt; 150K PKR monthly Household income</li> </ul> |
| Type of Tooth: [Mandibular 1 <sup>st</sup> Molar/ 2 <sup>nd</sup> Molar] |
| Side of the Tooth: [Right / Left] |
| Group Allocation: |
| Non-Ultrasonic Conventional Irrigation |
| <ul> <li>Ultrasonic Activated Irrigation.</li> </ul> |

# COMPARISION OF QUALITY OF OBTURATION AND LATERAL CANAL FILL (BY SEALER): ULTRASONIC ACTIVATED VERSUS NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUES IN ROOT CANAL TREATMENT:- A Randomized Controlled Trial

Dated: April 30, 2024

| Radiographic evaluation of obturation: | |
|---|---|
| Scoring | |
| - Length Score (0/1) | |
| - Density Score (0/1) | |
| - Taper Score (0/1) | |
| - Overall Obturation Quality Score (Sum of individual scores) | |
| Radiographic evaluation of Lateral canal Fill: | |
| Lateral canal filling (0/1) | |
| | Signature of Researcher |

COMPARISION OF QUALITY OF OBTURATION AND LATERAL CANAL FILL (BY SEALER): ULTRASONIC ACTIVATED VERSUS NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUES IN ROOT CANAL TREATMENT:-A Randomized Controlled Trial

Dated:April 30, 2024

Date: 30/04/2024

## **Inform consent form**

COMPARISION OF QUALITY OF OBTURATION AND LATERAL CANAL FILL (BY SEALER): ULTRASONIC ACTIVATED VERSUS NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUES IN ROOT CANAL TREATMENT:-A Randomized Controlled Trial

| Patient Name: |
|---|
| Father/ Husband Name: |
| I hereby, authorize concern doctor to include me in this study. The doctor has explained to me the |
| procedure of collection of data in detail and I fully understand that being part of this study sample |
| does not make me prone to any complications/ hazards. I have no binding or compulsion to be |
| part of this study and I have freedom to refuse from being part of this sample. |
| I have read this form and I am satisfied. |
| Name and signature of patient: |